CLINICAL TRIAL: NCT04930939
Title: Is Heart Rate Variability-guided Training Superior to Predefined Training for Improving Parasympathetic Activity and Aerobic Functional Capacity in Coronary Artery Disease Patients?
Brief Title: Heart Rate Variability-guided Training in Cardiac Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Manuel Moya, Principal investigator, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017.165.E.OEP
Record Dates: First submitted 2021-05-20; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Coronary Artery Disease
Keywords: Cardiorespiratory fitness; Cardiac vagal modulation; Heart rate variability; Cardiac rehabilitation
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Parallel assignment, two groups randomly assigned
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and assessors recoding the outcome measurements were blinded to the group allocations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heart rate variability-guided training group (Experimental): Patients allocated to heart rate variability-guided training group trained 3 days a week for 6 weeks. These patients carried out moderate continuous traininig sessions or high intensity interval training sessions based on their daily heart rate variability assessments follwing a decision schema.
  Interventions: Other: Aerobic training cardiac rehabilitation program
- Predefined training group (Active Comparator): Patients allocated to predefined training group also trained 3 days a week for 6 weeks. Nonetheless, these patients performed a predefined training program regarless of their parasympathetic modulation status.
  Interventions: Other: Aerobic training cardiac rehabilitation program

INTERVENTIONS:
Other: Aerobic training cardiac rehabilitation program — Moderate continuous training sessions and high intensity interval training sessiones were used to carried out aerobic training

SUMMARY:
Background: Previous studies have reported that heart rate variability (HRV)-guided training is a better option for improving autonomic function and aerobic capacity (i.e., oxygen uptake and power output at second ventilatory threshold and maximal exercise) during a cardiopulmonary exercise test compared to predefined training in sedentary and physically active healthy people. Nevertheless, none of these previous studies have been carried out with coronary artery disease (CAD) patients.

Methods: A total of 23 patients with CAD were divided into HRV-guided training group (HRV-G; n = 11) and predefined training group (PRE-G; n = 12). All patients trained three days a week for eight weeks (18 sessions). Patients allocated in the PRED-G carried out a previously established cardiac rehabilitation programme, combining sessions of moderate and high intensity, while patients allocated in the HRV-G carried out sessions of moderate or high intensity on the basis of their daily HRV assessments. The weekly averaged and isolated parasympathetic-related HRV indices, heart rate recovery, resting heart rate, and aerobic capacity were assessed before and after of the training programme.

DETAILED DESCRIPTION:
This study was a parallel-group, double-blind, randomised controlled trial. This study was approved by the ethical committee of the local University and was conducted conforming to the recommendations of the Declaration of Helsinki. Eligible patients were men and women with low-risk and age ≥ 18 years, who had experienced an acute myocardial infarction, angina pectoris, had undergone revascularisation (percutaneous transluminal coronary angioplasty or coronary artery bypass grafting) or coronary heart disease was documented by angiography, up to one year before to the enrolment in the study. Exclusion criteria included unstable angina, atrial fibrillation, cardiac implantable electronic devices, complex ventricular arrhythmias, uncontrolled hypertension, conditions limiting participation in exercise training and/or symptom-limited cardiopulmonary exercise test at pre-intervention. Before taking part in the study, patients were interviewed and signed a written informed consent. The patients were randomly allocated to a predefined training group (PRED-G; n = 12) or heart rate variability (HRV)-guided training group (HRV-G; n = 11).Before to start the study protocol, patients were instructed to properly carry out day-to-day HRV measurements. The study protocol was divided into two periods: a 2-week baseline period (BP) and a 6-week training period (TP). Before and after TP, baseline assessment week (PRE) and final assessment week (POST) were conducted, respectively. The variables/tests assessed/included in the assessment weeks were: cardiopulmonary exercise test, autonomic function, body composition, blood analysis, quality of life and dietary intake. Assessments were carried out in the same sequence and at the same period of the day. Patients and assessors recording the outcome measurements were blinded to the group allocations. Throughout the 6-week TP, patients allocated to PRED-G carried out a predefined training program, while patients that were assigned to HRV-G trained based on day-to-day HRV measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had experienced an acute myocardial infarction up to one year before to the enrolment in the study
* Patients who had experienced an angina pectoris up to one year before to the enrolment in the study
* Patients who had undergone revascularisation (percutaneous transluminal coronary angioplasty or coronary artery bypass grafting), up to one year before to the enrolment in the study
* Clinical diagnosis of coronary heart disease documented by angiography, up to one year before to the enrolment in the study

Exclusion Criteria:

* Unstable angina
* Atrial fibrillation
* Cardiac implantable electronic devices
* Complex ventricular arrhythmias
* Uncontrolled hypertension
* Conditions limiting participation in exercise training
* Symptom-limited cardiopulmonary exercise test at PRE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-12-23 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Change from PRE in workload at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), at the same period of the day
  A cardiopulmonary exercise test was performed using a medically supervised maximal graded cycle ergometer exercise test (Excite Bike Med, Technogym, Cesana, Italy) at the Miguel Hernandez University of Elche (Spain). The workload was obtained in Watts at the exercise peak and second ventilatory threshold. An experienced exercise physiologist together with a cardiologist supervised all the cardiorespiratory tests.
Change from PRE in absolute oxygen uptake at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), at the same period of the day
  A cardiopulmonary exercise test was performed using a medically supervised maximal graded cycle ergometer exercise test (Excite Bike Med, Technogym, Cesana, Italy) at the Miguel Hernandez University of Elche (Spain). Respiratory gas exchange was measured by MasterScreen CPX (Jaeger, Hoechberg, Germany). The oxygen uptake (VO2), expressed in absolute values (mL/min), was obtained at exercise peak, second ventilatory threshold and in resting condition. An experienced exercise physiologist together with a cardiologist supervised all the cardiorespiratory tests.
Change from PRE in relative oxygen uptake at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), at the same period of the day
  A cardiopulmonary exercise test was performed using a medically supervised maximal graded cycle ergometer exercise test (Excite Bike Med, Technogym, Cesana, Italy) at the Miguel Hernandez University of Elche (Spain). Respiratory gas exchange was measured by MasterScreen CPX (Jaeger, Hoechberg, Germany). The oxygen uptake (VO2), expressed in relative values to each individual's body weight (mL/kg/min), was obtained at exercise peak, second ventilatory threshold and in resting condition. An experienced exercise physiologist together with a cardiologist supervised all the cardiorespiratory tests.
Change from PRE in heart rate at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), at the same period of the day
  A cardiopulmonary exercise test was performed using a medically supervised maximal graded cycle ergometer exercise test (Excite Bike Med, Technogym, Cesana, Italy) at the Miguel Hernandez University of Elche (Spain). The heart rate (HR) was monitored continuously using a 12-lead electrocardiogram (Jaeger, Hoechberg, Germany). The HR was measured in beats per minute at exercise peak, second ventilatory threshold and in resting condition. An experienced exercise physiologist together with a cardiologist supervised all the cardiorespiratory tests.
Change from PRE in systolic blood pressure at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), at the same period of the day
  A cardiopulmonary exercise test was performed using a medically supervised maximal graded cycle ergometer exercise test (Excite Bike Med, Technogym, Cesana, Italy) at the Miguel Hernandez University of Elche (Spain). A digital sphygmomanometer (Tango+, Suntech, USA) was used for the assessment of systolic blood pressure. The systolic blood pressure was measured in millimetres of mercury at the exercise peak and in resting condition. An experienced exercise physiologist together with a cardiologist supervised all the cardiorespiratory tests.
Change from PRE in diastolic blood pressure at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), at the same period of the day
  A cardiopulmonary exercise test was performed using a medically supervised maximal graded cycle ergometer exercise test (Excite Bike Med, Technogym, Cesana, Italy) at the Miguel Hernandez University of Elche (Spain). A digital sphygmomanometer (Tango+, Suntech, USA) was used for the assessment of diastolic blood pressure. The diastolic blood pressure was measured in millimetres of mercury at the exercise peak and in resting condition. An experienced exercise physiologist together with a cardiologist supervised all the cardiorespiratory tests.
Change from PRE in isolated heart rate variability at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), at the same period of the day
  Isolated heart rate variability (HRV) assessments were performed in a quiet room with an average temperature of 22ᵒC. Polar H7 chest strap (Polar Electro OY, Kempele, Finland) and Elite HRV app (Perrotta, Jeklin, Hives, Meanwell, & Warburton, 2017) were used to capture HRV measurements. Patients were informed to avoid talking and sleeping, controlling breathing pace to 12 breaths per min. The length of the recording was 20 min, and the last 5 min was selected to calculate HRV indexes. Kubios HRV Software 2.0 for Windows (The Biomedical Signal Analysis Group, Kuopio, Finland) was used to analyse time and frequency domain indices in absolute and normalised units.
Change from PRE in averaged heart rate variability at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), after waking up
  All patients were instructed to assess their heart rate variability (HRV) in the morning at home every day throughout the entire study. The HRV recordings were attained via a photoplethysmography smartphone application (HRV4Ttraining) previously validated (Daniel J Plews et al., 2017). HRV assess were done at rest, as patients lay supine for 90 s with spontaneous breathing in a semi-dark room, and the las 60 s were capture. Day-to-day HRV values across assessment weeks (PRE and POST) were averaged to obtain a 7-day weekly averaged HRV value.
Change from PRE in heart rate recovery at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), at the same period of the day
  A cardiopulmonary exercise test was performed using a medically supervised maximal graded cycle ergometer exercise test (Excite Bike Med, Technogym, Cesana, Italy) at the Miguel Hernandez University of Elche (Spain). The heart rate (HR) was monitored continuously using a 12-lead electrocardiogram (Jaeger, Hoechberg, Germany). After the exercise peak, a 3-min cool-down at 10 W was performed. The reduction in HR from immediately exercise peak to the HR after 1 and 2 min was defined as HR recovery (HRR) 1 min and HRR 2 min, respectively. An experienced exercise physiologist together with a cardiologist supervised all the cardiorespiratory tests.

SECONDARY OUTCOMES:
Change from PRE in body mass index at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), at the same period of the day
  Body mass index (BMI) was calculated according to the formula: total weight in kilograms divided by squared height in meters (kg/m2). All anthropometrical variables were measured by a Level 2 anthropometrist certified by the International Society for the Advance of Kinanthropometry (ISAK).
Change from PRE in total body mass at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), at the same period of the day
  The total body mass of each participant was measured in kilograms using a digital scale (Tanita, TBF 300 A, Tokyo, Japan). All anthropometrical variables were measured by a Level 2 anthropometrist certified by the International Society for the Advance of Kinanthropometry (ISAK).
Change from PRE in breadths at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), at the same period of the day
  The breadths of each participant were measured with a Holtain bicondylar calliper (Holtain, UK). The following four breadths were measured: humerus, wrist, femur, and ankle. All anthropometrical variables were measured by a Level 2 anthropometrist certified by the International Society for the Advance of Kinanthropometry (ISAK).
Change from PRE in girths at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), at the same period of the day
  The total girths of each participant were measured with a metallic non-extensible tape (Lufkin, USA). The following four girths were measured: relaxed arm, flexed and tensed arm, thigh, and medial calf. All anthropometrical variables were measured by a Level 2 anthropometrist certified by the International Society for the Advance of Kinanthropometry (ISAK).
Change from PRE in skinfolds at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), at the same period of the day
  The skinfolds of each participant were measured with a Holtain Tanner/Whitehouse skinfold calliper (Holtain, UK). Eight skinfolds were also measured: triceps, biceps, subscapular, ileocrestal, supraspinale, abdominal, thigh, and medial calf. All anthropometrical variables were measured by a Level 2 anthropometrist certified by the International Society for the Advance of Kinanthropometry (ISAK).
Change from PRE in bone mass at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), at the same period of the day
  The percentage of bone mass of each participant was calculated according to Martin's equation. All anthropometrical variables were measured by a Level 2 anthropometrist certified by the International Society for the Advance of Kinanthropometry (ISAK).
Change from PRE in body fat mass at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), at the same period of the day
  The percentage of body fat mass of each participant was calculated using Durnin-Womersley equation. In addition, the sums of the eight skinfolds were considered for fat content calculations. All anthropometrical variables were measured by a Level 2 anthropometrist certified by the International Society for the Advance of Kinanthropometry (ISAK).
Change from PRE in muscle mass at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), at the same period of the day
  The percentage of muscle mass of each participant was calculated from Lee's equation. All anthropometrical variables were measured by a Level 2 anthropometrist certified by the International Society for the Advance of Kinanthropometry (ISAK).
Change from PRE in glucose at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), between 8:00 AM and 9:00 AM
  Blood samples were obtained from the median cubital vein at PRE and POST after at least a 10-hour fast and 48 h before the test and without performing exercise in that period. Venipuncture took place in the Vinalopó-Salud Hospital of Elche (Spain) and was carried out by a nurse. Glucose was measured using standard methods.
Change from PRE in urea at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), between 8:00 AM and 9:00 AM
  Blood samples were obtained from the median cubital vein at PRE and POST after at least a 10-hour fast and 48 h before the test and without performing exercise in that period. Venipuncture took place in the Vinalopó-Salud Hospital of Elche (Spain) and was carried out by a nurse. Urea was measured using standard methods.
Change from PRE in creatinine at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), between 8:00 AM and 9:00 AM
  Blood samples were obtained from the median cubital vein at PRE and POST after at least a 10-hour fast and 48 h before the test and without performing exercise in that period. Venipuncture took place in the Vinalopó-Salud Hospital of Elche (Spain) and was carried out by a nurse. Creatinine was measured using standard methods.
Change from PRE in uric acid at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), between 8:00 AM and 9:00 AM
  Blood samples were obtained from the median cubital vein at PRE and POST after at least a 10-hour fast and 48 h before the test and without performing exercise in that period. Venipuncture took place in the Vinalopó-Salud Hospital of Elche (Spain) and was carried out by a nurse. Uric acid was measured using standard methods.
Change from PRE in LDH at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), between 8:00 AM and 9:00 AM
  Blood samples were obtained from the median cubital vein at PRE and POST after at least a 10-hour fast and 48 h before the test and without performing exercise in that period. Venipuncture took place in the Vinalopó-Salud Hospital of Elche (Spain) and was carried out by a nurse. LDH was measured using standard methods.
Change from PRE in creatine kinase at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), between 8:00 AM and 9:00 AM
  Blood samples were obtained from the median cubital vein at PRE and POST after at least a 10-hour fast and 48 h before the test and without performing exercise in that period. Venipuncture took place in the Vinalopó-Salud Hospital of Elche (Spain) and was carried out by a nurse. Creatine kinase was measured using standard methods.
Change from PRE in sodium at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), between 8:00 AM and 9:00 AM
  Blood samples were obtained from the median cubital vein at PRE and POST after at least a 10-hour fast and 48 h before the test and without performing exercise in that period. Venipuncture took place in the Vinalopó-Salud Hospital of Elche (Spain) and was carried out by a nurse. Sodium was measured using standard methods.
Change from PRE in potassium at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), between 8:00 AM and 9:00 AM
  Blood samples were obtained from the median cubital vein at PRE and POST after at least a 10-hour fast and 48 h before the test and without performing exercise in that period. Venipuncture took place in the Vinalopó-Salud Hospital of Elche (Spain) and was carried out by a nurse. Potassium was measured using standard methods.
Change from PRE in cholesterol at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), between 8:00 AM and 9:00 AM
  Blood samples were obtained from the median cubital vein at PRE and POST after at least a 10-hour fast and 48 h before the test and without performing exercise in that period. Venipuncture took place in the Vinalopó-Salud Hospital of Elche (Spain) and was carried out by a nurse. Cholesterol was measured using standard methods.
Change from PRE in triglyerides at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), between 8:00 AM and 9:00 AM
  Blood samples were obtained from the median cubital vein at PRE and POST after at least a 10-hour fast and 48 h before the test and without performing exercise in that period. Venipuncture took place in the Vinalopó-Salud Hospital of Elche (Spain) and was carried out by a nurse. Triglycerides were measured using standard methods.
Change from PRE in HDL-C at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), between 8:00 AM and 9:00 AM
  Blood samples were obtained from the median cubital vein at PRE and POST after at least a 10-hour fast and 48 h before the test and without performing exercise in that period. Venipuncture took place in the Vinalopó-Salud Hospital of Elche (Spain) and was carried out by a nurse. HDL-C was measured using standard methods.
Change from PRE in LDL-C at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), between 8:00 AM and 9:00 AM
  Blood samples were obtained from the median cubital vein at PRE and POST after at least a 10-hour fast and 48 h before the test and without performing exercise in that period. Venipuncture took place in the Vinalopó-Salud Hospital of Elche (Spain) and was carried out by a nurse. LDL-C was measured using standard methods.
Change from PRE in haemoglobin A1c at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), between 8:00 AM and 9:00 AM
  Blood samples were obtained from the median cubital vein at PRE and POST after at least a 10-hour fast and 48 h before the test and without performing exercise in that period. Venipuncture took place in the Vinalopó-Salud Hospital of Elche (Spain) and was carried out by a nurse. Haemoglobin A1c was measured using standard methods.
Change from PRE in platelet at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), between 8:00 AM and 9:00 AM
  Blood samples were obtained from the median cubital vein at PRE and POST after at least a 10-hour fast and 48 h before the test and without performing exercise in that period. Venipuncture took place in the Vinalopó-Salud Hospital of Elche (Spain) and was carried out by a nurse. Platelet was measured using standard methods.
Change from PRE in red blood cells at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), between 8:00 AM and 9:00 AM
  Blood samples were obtained from the median cubital vein at PRE and POST after at least a 10-hour fast and 48 h before the test and without performing exercise in that period. Venipuncture took place in the Vinalopó-Salud Hospital of Elche (Spain) and was carried out by a nurse. Red blood cells were measured using standard methods.
Change from PRE in haemoglobin at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), between 8:00 AM and 9:00 AM
  Blood samples were obtained from the median cubital vein at PRE and POST after at least a 10-hour fast and 48 h before the test and without performing exercise in that period. Venipuncture took place in the Vinalopó-Salud Hospital of Elche (Spain) and was carried out by a nurse. Haemoglobin was measured using standard methods.
Change from PRE in quality of life at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), at the same period of the day
  The MacNew heart disease health-related quality of life (HRQL) instrument was used as a disease-specific health-related quality of life questionnaire. MacNew has been proved to be a valid and reliable questionnaire applicable to patients with coronary artery disease. The MacNew consists of 27 items that fall into three domains (a 13-item physical limitations domain scale, a 14-item emotional function domain scale, and a 13-item social function domain scale). The maximum possible score in any domain is 7 (high HRQL) and the minimum is 1 (poor HRQL).
Change from PRE in dietary intake at 6 weeks (POST) | Baseline (PRE) and at 6 weeks (POST), at the same period of the day
  Patients recorded food and beverage consumption during 4 consecutive days, including Sunday, before and after the intervention. Data from records were analyzed using the ST-Nutrition software (Servitux, Elche, Spain). Macro- and micronutrient intakes were evaluated paying attention to recommendations performed by the Portfolio dietary pattern for the National Cholesterol Education Program (NECP) Step II.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Miguel Hernández, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Undecided